CLINICAL TRIAL: NCT05942157
Title: Evaluation of the Efficacy and Safety of Antibiotic Therapeutic Drug Monitoring (TDM) in Patients With Difficult-to-Treat Gram-Negative Bacterial (DT-GNB) Infections
Brief Title: Therapeutic Drug Monitoring in Patients With Difficult-to-Treat Gram-Negative Bacterial Infections
Acronym: TDM-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDM RCT
Record Dates: First submitted 2023-06-20; First posted 2023-07-12 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Sepsis; Hemodynamic Instability; Bacterial Infections; Therapeutic Drug Monitoring; Antimicrobial Resistance
Keywords: Sepsis; Hemodynamic Instability; Therapeutic Drug Monitoring; Gram-negative Bacteria; Beta-Lactams; Fosfomycin; Fluoroquinolone; Glycylcycline; Dialysis
MeSH Terms: conditions — Sepsis; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The prescription of antibiotics will follow institution antibiotic prescribing guidelines or at the Infectious Disease (ID) clinician's discretion, based on culture and antibiotic susceptibilities results (whenever available). Empiric antibiotic treatment will be employed prior to the availability of culture or antibiotic susceptibilities results. Antibiotic level measurements, Minimum Inhibitory Concentrations (MIC) testing and Pharmacokinetics/Pharmacodynamics (PK/PD) target analysis will only be performed at Day 14 post enrolment, but the results will not be released to the ID clinician and the primary clinician.
- Intervention (Experimental): Once a positive GNB culture is known, antibiotic MIC testing will commence, and PK/PD target analysis will be performed using the antibiotic MIC. An every-other-day TDM-guided regimen will be chosen to rapidly adjust the antibiotic doses until the PK/PD target is achieved. In the event the antibiotic dose readjustment is unable to achieve the defined PK/PD target, blood sampling will continue every other day until Day 14 or the PK/PD target is achieved
  Interventions: Other: Therapeutic Drug Monitoring (TDM)

INTERVENTIONS:
Other: Therapeutic Drug Monitoring (TDM) — Upon randomization and before the bacterial culture results are known, blood sampling will be obtained from the patient during the morning round of initial empiric antibiotic administration. PK/PD target analysis based on the clinical susceptibility breakpoints of Enterobacterales (the most prevalent organism family of DT-GNB infections in our setting) will be performed and a dosage recommendation will be communicated to the primary ID clinician. Antibiotic dosing adjustments (if any) will be made within 8 - 24 hours of the blood sampling by the Primary / Infectious Diseases clinician. In case of inappropriate dosing, where the PK/PD target is not achieved or exceeded with antibiotic side effects observed, the dosage will be increased or decreased, respectively.
  Arms: Intervention

SUMMARY:
A prospective, open-label, randomized controlled trial will be conducted to evaluate a novel TDM-guided therapy in management of DT-GNB infections. We hypothesize that TDM-guided antibiotic therapy will reduce 14-day all-cause mortality by 6% (absolute risk reduction) in septic patients with DT-GNB infections, when compared to standard therapy. TDM for 11 antibiotics will be performed for all trial patients although test information will be withheld for the standard therapy arm. The primary aim is to compare the 14-day all-cause mortality rates of novel TDM-guided antibiotic dosing versus standard therapy.

DETAILED DESCRIPTION:
Sepsis remains a major cause of morbidity and mortality worldwide in the face of antimicrobial resistance especially in patients with Gram-negative bacteria (GNB) infections. Limited new antibiotics for GNB infections pose a severe threat to clinical management of these patients and thus call for old antibiotics to be repurposed. Dosing regimens of old antibiotics often fail to achieve therapeutic drug concentrations in some septic patients. Septic patients commonly have significant hemodynamic changes and/or undergo extracorporeal interventions that may increase patients' susceptibility to treatment failure and increase the chance of more resistant bacteria emergence, or toxicity from the antibiotic. Hence, the "one size fits all" dosing principle for antimicrobial treatments of suspect sepsis due to infection by antibiotic-resistant- or less susceptible-GNB [collectively known as "difficult-to-treat" (DT)-GNB infections] is no longer viable. This will require therapeutic drug monitoring (TDM) to inform if the dosing is adequate to treat such infections.

This study seeks to provide evidence supporting the application of TDM-guided antibiotic therapy on reducing mortality and morbidity among septic patients with DT-GNB infections and significant hemodynamic changes, which can potentially shift current practice paradigms.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Receive intravenous therapy of the study antibiotics
* Antibiotic treatment should be aimed for at least 3 days at time of inclusion

Exclusion Criteria:

* Pregnancy
* Antibiotics cessation before first blood sample collection
* Receiving antibiotics only as prophylaxis
* On palliative care or with less than 48 hours of life expectancy

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 810 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
14-day All-Cause Mortality Rate | 14 Days
  This is defined as death of any cause. Study aims to compare the difference in 14-day all-cause mortality rates from the day of randomization between both arms.

SECONDARY OUTCOMES:
Fever Resolution | 14 Days
  This is defined as the days to defervescence. Study aims to compare the difference in the days to defervescence after initiation of targeted antibiotic therapy between both arms.
Microbiological Treatment Cure of Difficult to Treat Gram-Negative Bacteria (DT-GNB) | 14 Days
  This is defined as presence of sterile site culture or absence of intended bacterial growth in culture of infection site. Study aims to compare microbiological cure of difficult to treat GNB between both arms.
Improved or Stabilized Sequential Organ Failure Assessment (SOFA) | 14 Days
  This is defined as delta SOFA or change in SOFA score between day 1 (randomization) to day 14. Study aims to compare the changes in SOFA scores between the two arms.
Incidences of Adverse Drug Reactions | Start to End of Antibiotic Therapy (Up to 90 days from randomization, discharge or demise, whichever comes earliest)
  Adverse Drug Reactions (ADRs) are defined as renal failure (defined using RIFLE criteria), Neurologic disorders (defined as altered mental status, peripheral neuropathy, or seizures in the absence of preexisting neurologic conditions, substance-related toxic effects, or infectious syndromes) and hematological disorders (defined as anemia (hemoglobin level <10 g/dL), leukopenia (white blood cell count <4500 cells/μL), or thrombocytopenia (platelet count <150 × 103/μL) with levels below patient's baseline and in the absence of bleeding or myelosuppressive therapies). Study aims to compare the incidences of ADRs between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Tze Peng Lim, PhD, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No